CLINICAL TRIAL: NCT07334210
Title: The Characteristics of Gut Microbiota in Patients With Sarcopenia and the Development of Probiotics
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Principal Investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2502-953-301
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia
Keywords: Gut microbiota; Sarcopenia; Older adults
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — oral microbiome and fecal microbiome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Sarcopenia patient group: Individuals aged 65 to 90 years.
  Meet the diagnostic criteria for sarcopenia based on the 2019 Asian Working Group for Sarcopenia (AWGS) guidelines:
  * Low appendicular skeletal muscle mass
    * DEXA: <7.0 kg/m² (men), <5.4 kg/m² (women)
    * BIA: <7.0 kg/m² (men), <5.7 kg/m² (women)
  * Low muscle strength
    * Handgrip strength: <28 kg (men), <18 kg (women) or
  * Low physical performance
    * 6-meter walk speed <1.0 m/s
    * 5-chair stand test ≥12 seconds
    * Short Physical Performance Battery (SPPB) score ≤9
- 2. Older adult control group: Individuals aged 65 to 90 years
- 3. Young adult control group: Individuals aged 20 to 50 years

SUMMARY:
The primary aim of this study is to identify the composition and characteristics of the gut microbiota in patients with sarcopenia in older adults, and compare these with the gut microbiota characteristics of older adults and young control groups to determine differences. Secondary purpose of this study is to provide data on the characteristics of gut microbiota for the development of probiotics effective in treating sarcopenia in older adults.

DETAILED DESCRIPTION:
Sarcopenia is a condition characterized by the loss of skeletal muscle mass and decline in physical function associated with aging. It is closely related to chronic diseases and geriatric disease and it is known to increase the risk of frailty, disability, falls, fractures, and mortality. The microbiome is closely associated with a wide range of human diseases, including metabolic disorders, cancer, infectious diseases, and immune-related conditions, and is considered one of the most valuable biomarkers for disease prevention and diagnosis. This indicates growing global interest and research activity on the connection between sarcopenia and gut microbiota. Through this study, we expect to elucidate the relationship between age-related sarcopenia and gut microbiota, which may provide important clues for the diagnosis and treatment of this condition.

ELIGIBILITY:
Inclusion criteria

1. Sarcopenia patient group

   * Individuals aged 65 to 90 years
   * Meet the diagnostic criteria for sarcopenia based on the 2019 Asian Working Group for Sarcopenia (AWGS) guidelines:
   * Low appendicular skeletal muscle mass

     * DEXA: <7.0 kg/m² (men), <5.4 kg/m² (women)
     * BIA: <7.0 kg/m² (men), <5.7 kg/m² (women)
   * Low muscle strength

     * Handgrip strength: <28 kg (men), <18 kg (women) or
   * Low physical performance

     * 6-meter walk speed <1.0 m/s
     * 5-chair stand test ≥12 seconds
     * Short Physical Performance Battery (SPPB) score ≤9
   * Voluntarily agree to participate in the clinical study and sign the informed consent form
2. Older adult control group

   * Individuals aged 65 to 90 years
   * Voluntarily agree to participate in the clinical study and sign the informed consent form
3. Young adult control group

   * Individuals aged 20 to 50 years
   * Voluntarily agree to participate in the clinical study and sign the informed consent form

Exclusion criteria

* Individuals currently under treatment for severe diseases of the cardiovascular, immune, respiratory, gastrointestinal/hepatic and biliary, renal/urinary, neurological, psychiatric systems, infectious diseases, or malignant tumors (Exception: skin tumors other than melanoma are excluded; cancer survivors may participate if more than 5 years have passed since complete remission).
* Individuals who have difficulty performing independent activities of daily living due to musculoskeletal or neurological diseases, or cognitive impairment (e.g., those with spinal disorders requiring surgery or having walking limitations).
* Individuals who regularly consume alcohol according to WHO daily intake standards (≥ 40 g/day for men, ≥ 20 g/day for women).
* Heavy smokers (≥ 20 cigarettes/day).
* Individuals with AST (GOT) or ALT (GPT) levels ≥ 3 times the upper limit of normal established by the testing institution.
* Patients with uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, measured after the subject has rested for 10 minutes).
* Patients with uncontrolled diabetes mellitus (HbA1c > 7.0%).
* Individuals with TSH ≤ 0.1 μIU/mL or ≥ 10 μIU/mL.
* Individuals deemed unsuitable for other reasons at the discretion of the investigator.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary general hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity analysis values | Baseline (visit 1)
  Alpha diversity analysis values (Rarefaction and Boxplot) of gut microbiota in each group
Short Physical Performance Battery (SPPB) | Screening(Visit 0)
  Short Physical Performance Battery (SPPB) results for sarcopenia physical performance evaluation in each group

SECONDARY OUTCOMES:
Beta diversity analysis values | Baseline(Visit 1)
  Beta diversity analysis values of gut microbiota (PCoA plot)
Taxa plot | Baseline(Visit 1)
  Taxa plot (Relative abundance) analysis values
Handgrip strength | Screening(Visit 0)
  Handgrip strength
6-meter walking speed | Screening(Visit 0)
  6-meter walking speed
appendicular skeletal muscle mass | Screening(Visit 0)
  appendicular skeletal muscle mass
lower limb muscle strength | Baseline (Visit 1)
  lower limb muscle strength
Timed Up & Go test | Baseline (Visit 1)
  Timed Up & Go test

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Young Lim, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No